CLINICAL TRIAL: NCT06988293
Title: The Evaluation of the Long-Term Quality of Life Effects of Laparoscopic Totally Extraperitoneal (TEP) and Lichtenstein Surgery in Inguinal Hernia Treatment
Brief Title: Quality of Life Effects of Laparoscopic and Open Surgery in Inguinal Hernia Treatment
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Ali Isler, Assistant Proffessor, Kahramanmaras Sutcu Imam University
Other Study IDs: KahramanmaraşSIU-İŞLER-001
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-01

CONDITIONS: İnguinal Hernia
Keywords: inguinal hernia, short form-36, total extraperitoneal(TEP) hernia repair, Liechtenstein hernia repair
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Liechtenstein and TEP hernia repair group
  Interventions: Procedure: inguinal hernia repair

INTERVENTIONS:
Procedure: inguinal hernia repair — İnguinal hernia repair quality of life index

SUMMARY:
Inguinal hernia is the most common type of hernia, presenting with swelling and pain in the groin area as clinical signs of abdominal wall hernias. The gold standard treatment for symptomatic inguinal hernias is surgery. There are various surgical methods for inguinal hernia repair. Tissue repair techniques such as Bassini, Shouldice, and McVay are no longer preferred due to their high recurrence rates, except in cases where mesh prosthetics are contraindicated. Tension-free mesh prosthesis-based anterior repairs and laparoscopic posterior repairs are the most frequently preferred methods in treatment. (1) In our study, we aimed to evaluate the quality of life index following laparoscopic extraperitoneal hernia repair using the most commonly preferred Lichtenstein technique. (2,3) The Short Form-36 (SF-36) scale is planned to be used for evaluating the quality of life index. SF-36 is one of the most commonly used generic measures for assessing quality of life. This scale examines eight dimensions of health, including physical function, social function, mental health, vitality (energy), pain, and general health perception, through 36 items. (4) Our study aims to determine which surgical method, based on long-term patient follow-up, stands out in improving the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* open and laparoscopic hernia repair surgery being over 18 years old approve the work

Exclusion Criteria:

* Being under 18 years old Emergency operated patients Patients using surgical techniques other than the open Liechtenstein method and laparoscopic extraperitoneal methods Patients who do not consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who had liechtenstein or TEP surgery due to inguinal hernia
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
SF-36 index | at least 1 year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü İmam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No